CLINICAL TRIAL: NCT00804960
Title: Controlled Ovarian Stimulation With Letrozole Supplementation
Brief Title: Does Letrozole Improve the Outcomes and/or Reduce the Cost of IVF-ET Cycles?
Acronym: Cost-Less
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of recruitment at this site
Sponsor: Center for Human Reproduction (Other)
Responsible Party: Kutluk Oktay, MD, Center for Human Reproduction
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHR #5/17/08-2
Record Dates: First submitted 2008-12-05; First posted 2008-12-09 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Infertility
Keywords: Cost of Infertility Treatment; Ovulation Induction; Letrozole; In Vitro Fertilization
MeSH Terms: conditions — Infertility | interventions — Letrozole; Ovulation Induction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Letrozole (Experimental): 1) Letrozole/ Recombinant FSH
  Interventions: Drug: Letrozole
- Standard IVF (Active Comparator): luteal phase GnRHa suppression/gonadotropin
  Interventions: Drug: Std IVF Protocol

INTERVENTIONS:
Drug: Letrozole — 1) Letrozole 5 mg starting on cycle day 2, which will be continued until the day of trigger. Recombinant FSH at doses 100-225 units, as determined by BMI, AFC, age, and ovarian reserve markers will be added on cycle day 4. The dose will be adjusted based on the response. An antagonist will be administered once the lead follicle reaches 14-mm in diameter or when estradiol level reaches 250 pg/mL. Oocyte maturation will be triggered by 20 iu of leuprolide acetate.
  Other Names: Femara
  Arms: Letrozole
Drug: Std IVF Protocol — 2) Long protocol with luteal phase GnRHa suppression with gonadotropin dose at 200-450 IU. Oocyte maturation will be triggered by 250 micg of ovidrel.
  Other Names: Ovulation induction with Human Menopausal gonoadotropins
  Arms: Standard IVF

SUMMARY:
This research is being done to determine whether the success rate of in vitro fertilization treatment can be improved, while lowering the cost incurred from infertility medications using a pill called letrozole.

DETAILED DESCRIPTION:
Specific Aim:

1. To determine whether addition of letrozole to gonadotropins would reduce the amount of gonadotropins used in an IVF-ET cycle, thereby reducing the cost.
2. To determine whether letrozole improves IVF-ET success compared to standard ovarian stimulation protocols.

Null Hypothesis: Use of Letrozole for ovulation induction in IVF is not less expensive than the standard therapy by a clinically relevant amount.

Alternative Hypothesis: Use of Letrozole for ovulation induction in IVF is better than the standard therapy by a clinically relevant amount.

Protocol:

Infertile women <40 years of age with age-appropriate ovarian reserve (as determined by day2/3 E2, FSH, and AMH) will be randomized between two protocols: one with letrozole and one with standard ovulation induction.

In both groups, serum FSH will be measured each time a sample is obtained for estradiol. Sera will be frozen for further batch assay.

Number of embryos to be transferred will be decided following the ASRM guidelines. The day of embryo transfer (D-3 vs D-5) will be based on the number and quality of embryos as per established clinical criteria.

Power Considerations

A review of 1473 cycles of patients less than 40 years old over the last 6 years (2002 - 2008) revealed average cost per cycle to be $3,152 +/- 1685(SD).

For the purpose of this power analysis we consider a 20% decrease in medication cost to be clinically significant. Thus a decrease from $ 3152.83 to $ 2522.26 will be considered clinically significant (20% decrease). For an alpha of 0.05 and a power of 80% for a two tailed test 113 patients will need to complete each arm.

Allowing for 10% drop-out we will attempt to randomize 125 patients to each arm of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Normal Ovarian Function
2. Normal uterus

Exclusion Criteria:

1. Age 40 and above
2. Diminished ovarian reserve (based on markers and/or previous poor response)
3. Previous oophorectomy

Ages: 21 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2009-12 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Cost of Treatment | 4 weeks

SECONDARY OUTCOMES:
Pregnancy and implantation rates | 4 weeks
Incidence of Ovarian Hyper stimulation Syndrome | 4 weeks
Multiple Birth Rate | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: David Barad, MD. MS, Study Director — CHR; Kutluk Oktay, MD, Principal Investigator — CHR/ New York Medical College
Locations (1):
- Center for Human Reproduction, New York, New York, United States